CLINICAL TRIAL: NCT03936114
Title: Stress Management and Resiliency Training (SMART) for Family Medicine Residents at Eglin AFB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Rhaney (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Laura Rhaney, Principal Investigator, Eglin AFB Regional Hospital
Organization: Eglin AFB Regional Hospital (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FWH20190021H
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Stress; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART (Experimental)
  Interventions: Behavioral: SMART

INTERVENTIONS:
Behavioral: SMART — SMART program mindfulness training program

SUMMARY:
This research seeks to identify if the practice of the SMART program mindfulness decreases stress and increase resilience in family medicine residents.

DETAILED DESCRIPTION:
This research seeks to identify if the practice of the SMART program mindfulness decreases stress and increase resilience in family medicine residents.

ELIGIBILITY:
**Patients must be able to get care at Eglin Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Male and female active duty military family medicine residents
* Age 18 or older
* Amenable to participation in training and filling out questionnaires

Exclusion Criteria:

* Unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Change in "Mindful Attention Awareness Scale" | baseline, 12 weeks, 12 months
  Dispositional mindfulness, i.e. open or receptive awareness of and attention to what is taking place in the present. To score the scale, compute a mean of the 15 questions. Higher scores reflect higher levels of dispositional mindfulness.
Change in "Perceived Stress Scale" | baseline, 12 weeks, 12 months
  The Perceived Stress Scale (PSS) is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. The PSS was designed for use in community samples with at least a junior high school education. The items are easy to understand, and the response alternatives are simple to grasp. Moreover, the questions are of a general nature and hence are relatively free of content specific to any subpopulation group. The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way. High scores indicate higher perceived stress.
Change in "Connor-Davidson Resilience Scale 10" (CD-RISC-10) | baseline, 12 weeks, 12 months
  Measure of stress coping ability. 10 questions with the option of 0 through 4, where 0 is not true at all and 4 is true nearly all the time. Scores are added up to obtain CD-RISC score.

CONTACTS AND LOCATIONS:
Locations (1):
- 96th Medical Group, Eglin Air Force Base, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data

REFERENCES:
- [Background] Ludwig DS, Kabat-Zinn J. Mindfulness in medicine. JAMA. 2008 Sep 17;300(11):1350-2. doi: 10.1001/jama.300.11.1350. No abstract available. PMID 18799450
- [Background] Holzel BK, Carmody J, Vangel M, Congleton C, Yerramsetti SM, Gard T, Lazar SW. Mindfulness practice leads to increases in regional brain gray matter density. Psychiatry Res. 2011 Jan 30;191(1):36-43. doi: 10.1016/j.pscychresns.2010.08.006. Epub 2010 Nov 10. PMID 21071182
- [Background] Kerr CE, Sacchet MD, Lazar SW, Moore CI, Jones SR. Mindfulness starts with the body: somatosensory attention and top-down modulation of cortical alpha rhythms in mindfulness meditation. Front Hum Neurosci. 2013 Feb 13;7:12. doi: 10.3389/fnhum.2013.00012. eCollection 2013. PMID 23408771
- [Background] Sibinga EM, Wu AW. Clinician mindfulness and patient safety. JAMA. 2010 Dec 8;304(22):2532-3. doi: 10.1001/jama.2010.1817. No abstract available. PMID 21139116
- [Background] Sood, Amit. Train Your Brain....Engage Your Heart....Transform Your Life: A Course in Attention & Interpretation Therapy (AIT). Morning Dew Publications, LLC; 2009, 2010

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT03936114/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT03936114/ICF_001.pdf